CLINICAL TRIAL: NCT02402959
Title: Individualized Treatment With Traditional Chinese Medicine Pattern Differentiation for the Patients With Insomnia Disorder: a Cohort Study
Brief Title: Individualized Treatment With Traditional Chinese Medicine for the Patients With Insomnia Disorder: a Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Baoyan Liu, vice-president, China Academy of Chinese Medical Sciences
Other Study IDs: GZR81230086
Record Dates: First submitted 2015-03-20; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Insomnia; Traditional Chinese Medicine; herbal medicine; cohort study; individualized treatment; TCM pattern differentiation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (10):
- Cohort 1: Based on the first TCM expert's experience and his knowledge, the insomnia patients will be treated with the best individualized treatment options, which should be at least in accordance to the current China Traditional Chinese herbal medicine pharmacopoeia and the China adult insomnia diagnosis and treatment guidelines. In addition, the expert could determine the treatment in consideration of individual patient's preferences and best existed evidence. Therefore, the choices of medicine, dosage form, dosage, frequency and duration are not restricted.
  Interventions: Other: individualized treatment
- Cohort 2: Based on the second TCM expert's experience and his knowledge, the insomnia patients will be treated with the best individualized treatment options, which should be at least in accordance to the current China Traditional Chinese herbal medicine pharmacopoeia and the China adult insomnia diagnosis and treatment guidelines. In addition, the expert could determine the treatment in consideration of individual patient's preferences and best existed evidence. Therefore, the choices of medicine, dosage form, dosage, frequency and duration are not restricted.
  Interventions: Other: individualized treatment
- Cohort 3: Based on the third TCM expert's experience and his knowledge, the insomnia patients will be treated with the best individualized treatment options, which should be at least in accordance to the current China Traditional Chinese herbal medicine pharmacopoeia and the China adult insomnia diagnosis and treatment guidelines. In addition, the expert could determine the treatment in consideration of individual patient's preferences and best existed evidence. Therefore, the choices of medicine, dosage form, dosage, frequency and duration are not restricted.
  Interventions: Other: individualized treatment
- Cohort 4: Based on the fourth TCM expert's experience and his knowledge, the insomnia patients will be treated with the best individualized treatment options, which should be at least in accordance to the current China Traditional Chinese herbal medicine pharmacopoeia and the China adult insomnia diagnosis and treatment guidelines. In addition, the expert could determine the treatment in consideration of individual patient's preferences and best existed evidence. Therefore, the choices of medicine, dosage form, dosage, frequency and duration are not restricted.
  Interventions: Other: individualized treatment
- Cohort 5: Based on the fifth TCM expert's experience and his knowledge, the insomnia patients will be treated with the best individualized treatment options, which should be at least in accordance to the current China Traditional Chinese herbal medicine pharmacopoeia and the China adult insomnia diagnosis and treatment guidelines. In addition, the expert could determine the treatment in consideration of individual patient's preferences and best existed evidence. Therefore, the choices of medicine, dosage form, dosage, frequency and duration are not restricted.
  Interventions: Other: individualized treatment
- Cohort 6: Based on the sixth TCM expert's experience and his knowledge, the insomnia patients will be treated with the best individualized treatment options, which should be at least in accordance to the current China Traditional Chinese herbal medicine pharmacopoeia and the China adult insomnia diagnosis and treatment guidelines. In addition, the expert could determine the treatment in consideration of individual patient's preferences and best existed evidence. Therefore, the choices of medicine, dosage form, dosage, frequency and duration are not restricted.
  Interventions: Other: individualized treatment
- Cohort 7: Based on the seven TCM expert's experience and his knowledge, the insomnia patients will be treated with the best individualized treatment options, which should be at least in accordance to the current China Traditional Chinese herbal medicine pharmacopoeia and the China adult insomnia diagnosis and treatment guidelines. In addition, the expert could determine the treatment in consideration of individual patient's preferences and best existed evidence. Therefore, the choices of medicine, dosage form, dosage, frequency and duration are not restricted.
  Interventions: Other: individualized treatment
- Cohort 8: Based on the eighth TCM expert's experience and his knowledge, the insomnia patients will be treated with the best individualized treatment options, which should be at least in accordance to the current China Traditional Chinese herbal medicine pharmacopoeia and the China adult insomnia diagnosis and treatment guidelines. In addition, the expert could determine the treatment in consideration of individual patient's preferences and best existed evidence. Therefore, the choices of medicine, dosage form, dosage, frequency and duration are not restricted.
  Interventions: Other: individualized treatment
- Cohort 9: Based on the nineth TCM expert's experience and his knowledge, the insomnia patients will be treated with the best individualized treatment options, which should be at least in accordance to the current China Traditional Chinese herbal medicine pharmacopoeia and the China adult insomnia diagnosis and treatment guidelines. In addition, the expert could determine the treatment in consideration of individual patient's preferences and best existed evidence. Therefore, the choices of medicine, dosage form, dosage, frequency and duration are not restricted.
  Interventions: Other: individualized treatment
- Cohort 10: Based on the tenth TCM expert's experience and his knowledge, the insomnia patients will be treated with the best individualized treatment options, which should be at least in accordance to the current China Traditional Chinese herbal medicine pharmacopoeia and the China adult insomnia diagnosis and treatment guidelines. In addition, the expert could determine the treatment in consideration of individual patient's preferences and best existed evidence. Therefore, the choices of medicine, dosage form, dosage, frequency and duration are not restricted.
  Interventions: Other: individualized treatment

INTERVENTIONS:
Other: individualized treatment — Individualized treatment includes anything no matter what kind of interventions, like medicine, herbs, acupuncture, massage, behaviour therapy, diet and exercise therapy. The TCM experts should choose the intervention in accordance to the patients' preference, best existed evidence and their empirical knowledge.

SUMMARY:
The primary purpose of this study is to discover, establish and refine the individual treatment protocol of each TCM expert for insomnia, and to explore what characteristics of the patients are considered with the corresponding treatment in clinical practices.

The secondary purpose is to determine the effectiveness of TCM pattern differentiation treatment for the patients with insomnia.

DETAILED DESCRIPTION:
Traditional Chinese medicine (TCM) has been effectively and instantly used for keeping Chinese people's health over 2000 years. Recently the TCM is becoming popular and well known home and abroad due to its effectiveness and individualized treatment. It has been known that TCM practitioners diagnosed, give the treatment and evaluated patients' health condition with symptoms and signs, what are called TCM patterns. This is why TCM practitioners always consider and emphasize the importance of TCM patterns in the TCM education and clinic practices. At the same time, TCM pattern differentiation is considered complicated and difficult to understand, due to the difference of TCM practitioners'clincal experience and knowledge. The one ,who has more experience and knowledge, treat patients more effective than the other. Unlike modernized medicine, drugs are not always recommended for the diseases, conversely, the TCM practitioners and their knowledge are always recommended. In addition, young TCM practitioners have to follow and imitate the experts who are full of knowledge, if they want to be good ones. From these views, the experience and knowledge of experts are important and crucial to the clinical outcomes, meanwhile they are hard to discover and establish. Therefore, we package the experts and their treatment as the one target to discover, establish and refine the individual treatment protocol (experience and knowledge) of each TCM expert, and to explore what characteristics of the patients are considered with the corresponding treatment in clinical practices.

The prerequisite of the study is that experts chosen for the study are the ones who are the specialists on the insomnia treatment. So, the secondary purpose is to determine the effectiveness of TCM patter differentiation treatment for the patients with insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the diagnosis of insomnia;
2. Patients' age between 18 and 65 years (18 and 65 years included);
3. Patients with the oral or written informed consent.

Exclusion Criteria:

1. Patients with any uncontrolled and severe diseases which cause insomnia will be excluded. the diseases may include heart disease (like angina, cardiac arrhythmias, heart failure, myocardial infarction), pulmonary disease (COPD, asthma), gastrointestinal disorders (stomach or duodenal ulcers, reflux disease), neurologic disorders (seizures, spastic torticollis, blepharospasm, dystonias, parkinson's disease, alzheimer's disease, dementia, sleep-disruptive headaches), head trauma (blow to the head with loss of consciousness, concussion), pain disorders (fibrositis/fibromyalgia, arthritis, muscle cramps, chronic low back pain, headaches), endocrine and metabolic disorders (thyroid disease, diabetes), kidney disease (kidney failure with dialysis, kidney stones) autoimmune disorders, cancer, and HIV/AIDS.
2. Psychopath with suicidal tendency;
3. Patients with pregnancy and lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnosis of insomnia, who come to the experts' clinic for treatment, will be invitated and included in his cohort.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Sleep Quality | Week 1, 2, 4, 6, 8 or Final visit.
  Measured by Pittsburgh Sleep Quality Index, PSQI

SECONDARY OUTCOMES:
Change from baseline in the diagnosis of insomnia | Week 1, 2, 4, 6, 8 or Final visit.
  Measured by the Structured Interview for Insomnia Disorder (SID), which is a translation and modified version of Brief Insomnia Questionnaire and used as a diagnosis questionnaire in the study. Its content validity has been reviewed and assessed by the experts who participated in the cohort. Three criteria of DSM-Ⅴ, ICSD-3 and ICD-10 for insomnia have been included in the SID questionnaire. The SID is chosen as an outcome to tell whether there is a diagnosis of insomnia after treatment.
Change from baseline in the Insomnia Severity | Week 1, 2, 4, 6, 8 or Final visit.
  Measured by Insomnia Severity Index, ISI
Change from baseline in the Patient's satisfaction to the TCM treatment | Week 1, 2, 4, 6, 8 or Final visit.
  Measured by the Patient's satisfaction scale
Change from baseline in the Insomnia severity and improvement | Week 1, 2, 4, 6, 8 or Final visit.
  Measured by the Clinician Global Impression Scale-Severity and -Improvement score.
Change from baseline in the Clinician's satisfaction to the TCM treatment | Week 1, 2, 4, 6, 8 or Final visit.
  Measured by the Clinician Reported Outcome for TCM treatment
Change from baseline in the Reduction of western medicine | Week 1, 2, 4, 6, 8 or Final visit.
  Reported by the patients.
Change from baseline in the Sleep structure | Week 1, 2, 4, 6, 8 or Final visit.
  Measured by the Cardiopulmonary Coupling (CPC), which is a new operator-independent, automated measure of sleep physiology. CPC collects the electrocortical activity of the heart rate variability (HRV) and respiration. The result provides information on sleep quality and sleep disordered breathing phenotypes independent of EEG analysis. High-frequency coupling states the consolidated and stable NREM sleep, and Low-frequency coupling is enhanced in states of fragmented sleep.
Change from baseline in the Depression/Anxiety severity | Week 1, 2, 4, 6, 8 or Final visit.
  Measured by the Hamilton Depression/Anxiety Scale
Change from baseline in the Other measures that experts regard them necessary. | Week 1, 2, 4, 6, 8 or Final visit.
  Other measures may include the wrist actigraphy, Polysomnography (PSG), other questionnaires, Multiple Sleep Latency Test (MSLT), CT, MRI, or some chemicals test.
Adverse Event | Week 1, 2, 4, 6, 8 or Final visit.
  Reported by the patients, such as cold, fever, diarrhea, and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Baoyan Liu, Master, Principal Investigator — China Academy of Chinese Medical Sciences
Locations (7):
- China (7):
  - East Hospital of Beijing University of Traditional Chinese Medicine, Beijing, Beijing Municipality
  - Guang'anmen Hospital of China Academy of China Medical Sciences, Beijing, Beijing Municipality
  - Fujian Institute of Traditional Chinese Medicine, Fuzhou, Fujian
  - Shenzhen hospital of Traditionl Chinese Medicine, Shenzhen, Guangdong
  - Affiliated hospital of He'nan university of Traditional Chinese Medicine, Zhengzhou, Henan
  - Clinic of Hubei university of Traditional Chinese Medicine, Wuhan, Hubei
  - Affiliated hospital of Shandong university of Traditional Chinese Medicine, Ji'nan, Shandong